CLINICAL TRIAL: NCT02771626
Title: A Phase 1/2 Study of the Safety, Pharmacokinetics, and Pharmacodynamics of the Glutaminase Inhibitor CB-839 in Combination With Nivolumab in Patients With Advanced/Metastatic Melanoma, Renal Cell Carcinoma and Non-Small Cell Lung Cancer
Brief Title: Study CB-839 in Combination With Nivolumab in Patients With Melanoma, Clear Cell Renal Cell Carcinoma (ccRCC) and Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-004
Record Dates: First submitted 2016-05-06; First posted 2016-05-13 (Estimated); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Clear Cell Renal Cell Carcinoma (ccRCC); Melanoma; Non-small Cell Lung Cancer (NSCLC)
Keywords: RCC; Melanoma (MEL); NSCLC; Immuno-Oncology; Tumor Metabolism; Glutaminase; Glutaminase Inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — CB-839; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Telaglenastat 600 mg + Standard Dose Nivolumab (Experimental): Telaglenastat 600 mg in combination with standard dose nivolumab in participants with advanced/metastatic clear cell renal cell carcinoma (ccRCC), melanoma, and non-small cell lung cancer (NSCLC).
  Interventions: Drug: CB-839; Drug: Nivolumab
- Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors (Experimental): Telaglenastat 800 mg/standard dose nivolumab combination in participants with advanced/metastatic ccRCC who have previously received at least one tyrosine kinase inhibitor (TKI) but are treatment naïve to checkpoint modulators programmed death-1/programmed death ligand-1 (PD-1/PD-L1), cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), or any other agent that specifically targets a T-cell checkpoint or co-stimulation pathway.
  Interventions: Drug: CB-839; Drug: Nivolumab
- Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab (Experimental): Telaglenastat 800 mg/standard dose nivolumab combination in participants with advanced/metastatic ccRCC who received nivolumab in most recent treatment line that had documented radiological disease progression OR are currently receiving nivolumab with stable disease for at least 24 weeks.
  Interventions: Drug: CB-839; Drug: Nivolumab
- Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy (Experimental): Telaglenastat 800 mg/standard dose nivolumab combination in participants with advanced/metastatic ccRCC that had documented radiological disease progression while receiving an anti-PD-1/PD-L1 therapy in any prior line of therapy.
  Interventions: Drug: CB-839; Drug: Nivolumab
- Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy (Experimental): Telaglenastat 800 mg/standard dose nivolumab combination in participants with unresectable or metastatic melanoma that had documented radiological disease progression while receiving an anti-PD-1 therapy in their most recent line of therapy.
  Interventions: Drug: CB-839; Drug: Nivolumab
- Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy (Experimental): Telaglenastat 800 mg/standard dose nivolumab combination in participants with NSCLC that does not harbor an activating mutation in the epidermal growth factor receptor (EGFR) oncogene and who received nivolumab in most recent treatment line and had documented radiological disease progression OR are currently receiving nivolumab with Stable Disease for at least 24 weeks.
  Interventions: Drug: CB-839; Drug: Nivolumab

INTERVENTIONS:
Drug: CB-839 — Glutaminase inhibitor
  Other Names: telaglenastat
Drug: Nivolumab — PD-1 inhibitor
  Other Names: Opdivo; BMS-936558

SUMMARY:
This study is an open-label Phase 1/2 evaluation of CB-839 in combination with nivolumab in participants with clear cell renal cell carcinoma, melanoma, and non-small cell lung cancer.

ELIGIBILITY:
Addition eligibility criteria based on tumor type apply

Inclusion Criteria:

* Ability to provide written informed consent in accordance with federal, local, and institutional guidelines
* Histological or cytological diagnosis of metastatic cancer or locally advanced cancer that is not amenable to local therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life Expectancy of at least 3 months
* Adequate hepatic, renal, cardiac, and hematologic function
* Measurable disease by Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 criteria
* Resolution of treatment-related toxicities except alopecia

Exclusion Criteria:

* Unable to receive oral medications
* Unable to receive oral or intravenous (IV) hydration
* Intolerance to prior anti-PD-1/PD-L1 therapy
* Prior severe hypersensitivity reaction to another monoclonal antibody (mAb)
* Any other current or previous malignancy within 3 years except protocol allowed malignancies
* Chemotherapy, TKI therapy, radiation therapy or hormonal therapy within 2 weeks
* Immunotherapy or biological therapy, or investigational agent within 3 weeks (Note: Some cohort exceptions allow anti-PD-1 therapy)
* Active known or suspected exclusionary autoimmune disease
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other systemic immunosuppressive medications within 2 weeks
* History of known risks factors for bowel perforation
* Symptomatic ascites or pleural effusion
* Major surgery within 28 days before Cycle 1 Day 1
* Active infection requiring parenteral antibiotics, antivirals, or antifungals within 2 weeks prior to first dose of study drug
* Patients who have human immunodeficiency virus (HIV), Hepatitis B or C
* Conditions that could interfere with treatment or protocol-related procedures
* Active and/or untreated central nervous system (CNS) disease or non-stable brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Whiting, MD, PhD, Study Director — Calithera Biosciences, Inc
Locations (17):
- United States (17):
  - Honor Health, Scottsdale, Arizona
  - Stanford University, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - University Cancer Blood Center, Athens, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Caner Center, Detroit, Michigan
  - New York University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance/University of Washington, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
Started | 8 | 26 | 17 | 9 | 37 | 21
Completed (Study was terminated early. Participants still on study at the time of the study termination (see Reason Not Completed=Study Termination by Sponsor, below) were transferred to individual patient treatment Investigational New Drug applications (INDs) per physician and participant request.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 26 | 17 | 9 | 37 | 21
Not completed — Adverse Event | 1 | 5 | 3 | 0 | 1 | 1
Not completed — Radiologic Disease Progression | 6 | 13 | 10 | 7 | 28 | 15
Not completed — Symptomatic Deterioration | 0 | 4 | 2 | 0 | 5 | 2
Not completed — Participant Request | 0 | 1 | 0 | 2 | 0 | 1
Not completed — Investigator Decision | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Study Termination by Sponsor | 0 | 2 | 1 | 0 | 1 | 0
Not completed — Informed Consent Withdrawn | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Other, Not Specified | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Telaglenastat 600 mg + Standard Dose Nivolumab: Telaglenastat 600 mg in combination with standard dose nivolumab in participants with advanced/metastatic ccRCC, melanoma, and NSCLC.
- Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors: Telaglenastat 800 mg/standard dose nivolumab combination in participants with advanced/metastatic ccRCC who have previously received at least one TKI but are treatment naïve to checkpoint modulators PD-1/PD-L1, CTLA-4, or any other agent that specifically targets a T-cell checkpoint or co-stimulation pathway.
- Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy: Telaglenastat 800 mg/standard dose nivolumab combination in participants with NSCLC that does not harbor an activating mutation in the EGFR oncogene and who received nivolumab in most recent treatment line and had documented radiological disease progression OR are currently receiving nivolumab with Stable Disease for at least 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy | Total
Number analyzed (Participants) | 8 | 26 | 17 | 9 | 37 | 21 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (13.51) | 58.4 (10.75) | 67.8 (9.85) | 63.2 (7.90) | 63.4 (11.82) | 67.0 (11.55) | 63.3 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 3 | 2 | 15 | 11 | 42
  Male | 5 | 18 | 14 | 7 | 22 | 10 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 0 | 2 | 1 | 8
  Not Hispanic or Latino | 6 | 23 | 17 | 9 | 33 | 20 | 108
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 0 | 0 | 4 | 8
  White | 8 | 19 | 16 | 9 | 34 | 15 | 101
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Dose Interruption, Reduction, or Study Drug Discontinuation (Excluding Grade 5 Disease Progression)
Description: An adverse event (AE) is any untoward, undesired, or unplanned event that does not need to be causally related to treatment. A serious adverse event (SAE) is an AE that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in a persistent or significant disability or incapacity, results in a congenital anomaly or birth defect, or important medical events that may not result in death, be life-threatening, or require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Relatedness to study medication was graded as either, probably, possibly, unlikely, or unrelated. Events were categorized according to the Common Toxicity Criteria for Adverse Events (CTCAE) Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening, Grade 5=death.
Time Frame: From the first dose of study drug up to 28 days post last dose. Median duration of telaglenastat treatment was 92 days and that for nivolumab treatment was 84 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
Number analyzed (Participants) | 8 | 26 | 17 | 9 | 37 | 21
Participants
  ≥ 1 TEAE | 8 | 26 | 17 | 9 | 36 | 21
  ≥ 1 TEAE ≥ grade 3 | 5 | 17 | 8 | 4 | 17 | 12
  ≥ 1 TEAE related to nivolumab | 6 | 22 | 15 | 8 | 28 | 17
  ≥ 1 TEAE related to telaglenastat | 4 | 24 | 15 | 9 | 28 | 17
  ≥ 1 TEAE ≥ grade 3 related to nivolumab | 0 | 6 | 6 | 2 | 4 | 5
  ≥ 1 TEAE ≥ grade 3 related to telaglenastat | 0 | 5 | 6 | 2 | 4 | 4
  ≥ 1 grade 5 TEAE related to nivolumab | 0 | 0 | 0 | 0 | 0 | 0
  ≥ 1 grade 5 TEAE related to telaglenastat | 0 | 0 | 0 | 0 | 0 | 0
  ≥ 1 TEAE leading to discontinuation (DC) of nivolumab | 1 | 6 | 3 | 0 | 1 | 3
  ≥ 1 TEAE leading to DC of telaglenastat | 0 | 5 | 3 | 0 | 2 | 3
  ≥ 1 TEAE leading to DC of nivolumab and telaglenastat | 0 | 4 | 3 | 0 | 1 | 3
  ≥ 1 TEAE leading to DC of nivolumab or telaglenastat | 1 | 6 | 3 | 0 | 2 | 3
  ≥ 1 TEAE requiring nivolumab dose interruption or reduction | 4 | 15 | 10 | 6 | 9 | 5
  ≥ 1 TEAE requiring telaglenastat dose interruption or reduction | 4 | 16 | 9 | 6 | 14 | 10
  ≥ 1 TEAE requiring nivolumab and telaglenastat dose interruption or reduction | 3 | 15 | 9 | 4 | 8 | 5
  ≥ 1 TEAE requiring nivolumab or telaglenastat dose interruption or reduction | 4 | 16 | 10 | 8 | 15 | 10
  ≥ 1 grade 5 TEAE | 1 | 1 | 0 | 0 | 0 | 0
  ≥ 1 serious TEAE | 2 | 7 | 6 | 1 | 9 | 6
  ≥ 1 serious TEAE ≥ grade 3 | 1 | 6 | 5 | 1 | 8 | 4
  ≥ 1 serious TEAE related to nivolumab | 0 | 4 | 1 | 1 | 3 | 2
  ≥ 1 serious TEAE related to telaglenastat | 0 | 3 | 2 | 0 | 2 | 3
  ≥ 1 serious TEAE ≥ grade 3 related to nivolumab | 0 | 3 | 1 | 1 | 3 | 2
  ≥ 1 serious TEAE ≥ grade 3 related to telaglenastat | 0 | 2 | 2 | 0 | 2 | 3

2. Primary Outcome: Number of Participants With Clinically Significant Treatment-Emergent Values in Hematology, Serum Chemistry Panel, Vital Signs or Weight
Description: Hematology assessments included: hemoglobin; hematocrit, red blood cell count, white blood cell count with differential, and platelet count. Serum chemistry panel included: sodium, potassium, chloride, carbon dioxide, calcium, glucose, blood urea nitrogen, total protein, albumin, total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, lactate dehydrogenase, creatinine, thyroid stimulating hormone. Vital sign assessments included systolic and diastolic blood pressures, pulse (heart) rate, respiratory rate, temperature, and body weight.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
Number analyzed (Participants) | 8 | 26 | 17 | 9 | 37 | 21
Participants
  Hematology Values | 0 | 3 | 1 | 0 | 1 | 1
  Clinical Laboratory Values | 1 | 4 | 3 | 0 | 2 | 2
  Vital Sign Values | 0 | 0 | 0 | 0 | 0 | 0
  Weight | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Overall Response Rate (ORR) Per Investigator Assessed Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR or PR was required to be sustained for 4 weeks when confirmation was reported.
  * CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: up to a maximum of 2.8 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
Number analyzed (Participants) | 8 | 26 | 17 | 9 | 37 | 21
percentage of participants | 0 [0.0 to 36.9] | 24.0 [9.4 to 45.1] | 5.9 [0.1 to 28.7] | 0 [0 to 33.6] | 5.4 [0.7 to 18.2] | 0.0 [0.0 to 17.6]

4. Primary Outcome: Duration of Response (DOR) Per Investigator Assessed RECIST v1.1
Description: DOR is defined as the time between the first documentation of a PR or a CR to the first documentation of progressive disease (PD) or death, whichever occurred first. DOR was censored at the date of last radiographic disease if the patient was alive and progression free at the time of database lock, PD, or death occurred after missing data for 2 consecutive radiographic disease assessments, or patient received non-protocol treatment prior to documentation of disease progression.
  * CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: up to a maximum of 2.8 years
Population: Participants with a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
Number analyzed (Participants) | 0 | 6 | 1 | 0 | 2 | 0
months |  | 13.01 [11.01 to NA] — Upper limit of confidence interval not available due to insufficient events above the median. | 3.71 [NA to NA] — Not applicable since 1 participant analyzed. |  | 9.59 [4.53 to 14.65] |

5. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1
Description: PFS was defined as time from the first dose date to the earlier of either PD per RECIST v1.1 or death from any cause. The duration of PFS was censored at the date of last radiographic disease if the patient was alive and progression-free at the time of analysis data cutoff, disease progression, or death occurred after missing data for 2 consecutive radiographic disease assessments, or patient received non-protocol treatment prior to documentation of disease progression.
  - PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: up to a maximum of 2.8 years
Population: Participants with an event (PD per RECIST v1.1 or death from any cause).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
Number analyzed (Participants) | 8 | 18 | 14 | 7 | 32 | 17
months | 3.42 [1.74 to 9.33] | 3.72 [1.84 to 12.85] | 3.71 [1.87 to 5.52] | 1.87 [1.81 to 5.52] | 2.07 [1.87 to 3.75] | 2.20 [1.74 to 5.59]

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first dose date to death due to any cause. For participants alive at time of analysis, overall survival was censored at the time when the participant was last known to be alive.
Time Frame: up to a maximum of 2.8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
Number analyzed (Participants) | 8 | 26 | 17 | 9 | 37 | 21
months | NA [8.25 to NA] — Insufficient events to establish the median and upper confidence limit. | 24.54 [16.30 to NA] — Upper limit of confidence interval not available due to insufficient events above the median. | 22.57 [14.62 to NA] — Upper limit of confidence interval not available due to insufficient events above the median. | NA [26.25 to NA] — Insufficient events to establish the median and upper confidence limit. | 10.91 [8.87 to 18.14] | 8.61 [4.11 to 19.71]

ADVERSE EVENTS:
Time Frame: All Cause Mortality: up to a maximum of 2.8 years. Adverse Events: from the first dose of study drug up to 28 days post last dose. Median duration of telaglenastat treatment was 92 days and that for nivolumab treatment was 84 days.
Description: Per protocol, serious adverse events exclude those of Grade 5 disease progression.
Arm/Group | Telaglenastat 600 mg + Standard Dose Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy
All-Cause Mortality (participants affected / at risk) | 3/8 | 15/26 | 11/17 | 3/9 | 27/37 | 16/21
Serious Adverse Events (participants affected / at risk) | 2/8 | 8/26 | 6/17 | 1/9 | 12/37 | 7/21
Other Adverse Events (participants affected / at risk) | 8/8 | 26/26 | 15/17 | 9/9 | 36/37 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telaglenastat 600 mg + Standard Dose Nivolumab (N=8) | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors (N=26) | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab (N=17) | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy (N=9) | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy (N=37) | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy (N=21)
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Immune system disorder (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telaglenastat 600 mg + Standard Dose Nivolumab (N=8) | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Naïve to Checkpoint Inhibitors (N=26) | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC Recently Treated With Nivolumab (N=17) | Telaglenastat 800 mg + Standard Dose Nivolumab: ccRCC With Prior PD-1 Therapy (N=9) | Telaglenastat 800 mg + Standard Dose Nivolumab: Melanoma With Prior PD-1 Therapy (N=37) | Telaglenastat 800 mg + Standard Dose Nivolumab: NSCLC With Prior PD-1 Therapy (N=21)
Nausea (Gastrointestinal disorders) | 3 | 7 | 6 | 5 | 16 | 9
Constipation (Gastrointestinal disorders) | 1 | 5 | 5 | 4 | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 9 | 3 | 3 | 6 | 4
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3 | 2 | 6 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 1 | 0 | 8 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6 | 7 | 3 | 6 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5 | 4 | 1 | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 2 | 5 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 4 | 1
Fatigue (General disorders) | 2 | 14 | 8 | 6 | 12 | 8
Oedema peripheral (General disorders) | 2 | 6 | 2 | 0 | 3 | 2
Pain (General disorders) | 0 | 7 | 3 | 0 | 1 | 1
Chills (General disorders) | 1 | 2 | 3 | 1 | 3 | 0
Pyrexia (General disorders) | 0 | 2 | 2 | 1 | 3 | 2
Arthralgia (General disorders) | 4 | 7 | 3 | 1 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3 | 1 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2 | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 5 | 4 | 1 | 11 | 3
Alanine aminotransferase increased (Investigations) | 0 | 8 | 4 | 2 | 7 | 2
Blood creatinine increased (Investigations) | 2 | 5 | 4 | 1 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 3 | 1 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 4 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 2 | 1 | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8 | 4 | 4 | 3 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 4 | 3 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 2 | 3 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 2 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 2
Photophobia (Eye disorders) | 1 | 12 | 4 | 3 | 12 | 6
Vision blurred (Eye disorders) | 1 | 6 | 1 | 1 | 3 | 0
Visual impairment (Eye disorders) | 1 | 2 | 0 | 2 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 5 | 4 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1 | 1 | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 5 | 5 | 2 | 5 | 3
Dizziness (Nervous system disorders) | 0 | 4 | 3 | 2 | 7 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 4 | 2 | 8 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 5 | 2 | 1 | 4 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 5 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1 | 1 | 4
Hypotension (Vascular disorders) | 0 | 3 | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication by the PI before either a multi-site publication or 18 months after final multi-site study report. PI can only publish their own results and provide 45 days in advance notice. PI must delete any Calithera confidential information from the publication other than study results and give good faith consideration to other comments made by Calithera. The PI must delay the publication for up to 45 days if requested by Calithera and publicly acknowledge Calithera and Pfizer support.

DOCUMENTS (2):
  • Study Protocol (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT02771626/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT02771626/SAP_001.pdf